CLINICAL TRIAL: NCT02331745
Title: Granulocyte Colony-stimulating Factor(G-CSF) in the Treatment of Hepatic Failure: a Prospective Randomized Controlled Clinical Study
Brief Title: RCT Study on Granulocyte Colony-stimulating Factor(G-CSF) Treatment of Hepatic Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Jinhua Hu, Prof. & Chief Physician, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z131107002213157
Record Dates: First submitted 2014-12-24; First posted 2015-01-06 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Liver Failure; Hepatitis B; Alcoholic Liver Disease
MeSH Terms: conditions — Liver Failure; Hepatitis B; Liver Diseases, Alcoholic | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Granulocyte colony-stimulating factor (Experimental): Granulocyte colony-stimulating factor(G-CSF) was given 5 ug/kg subcutaneously qd for 6 doses,then qod for other 6 doses(total 12 doses).
  Standard treatment includes reduced glutathione, glycyrrhizin, ademetionine,polyene phosphatidylcholine, alprostadil, and human serum albumin) on the day of admission. HBV associated ACLF patients receive entecavir at the same time
  Interventions: Drug: Granulocyte colony-stimulating factor; Drug: standard treatment
- standard treatment (Active Comparator): Standard treatment alone
  Interventions: Drug: standard treatment

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor — Granulocyte colony-stimulating factor(G-CSF) was given 5 ug/kg subcutaneously qd for 6 doses,then qod for other 6 doses(total 12 doses).
  Other Names: G-CSF
  Arms: Granulocyte colony-stimulating factor
Drug: standard treatment — Standard treatment includes reduced glutathione, glycyrrhizin, ademetionine,polyene phosphatidylcholine, alprostadil, and human serum albumin) on the day of admission. HBV associated ACLF patients receive entecavir at the same time
  Other Names: SDT

SUMMARY:
This study evaluates the Granulocyte colony-stimulating factor (G-CSF) in the treatment of Acute on Chronic Liver Failure in adult. Half participants will receive G-CSF and standard treatment in combination, while half participants will receive standard treatment.

DETAILED DESCRIPTION:
Granulocyte colony-stimulating factor (G-CSF) can be used to mobilize stem cells to the periphery and the liver tissue in patients with advanced liver disease, and could promote hepatic regeneration. Moreover, G-CSF was reported to protect patients from sepsis by restoring the function of both neutrophils and monocytes. Therefore, G-CSF therapy may be beneficial for liver regeneration in patients with ACLF induced by different causes.

standard therapy for the treatment of ACLF includes reduced glutathione, glycyrrhizin, ademetionine,polyene phosphatidylcholine, alprostadil, and human serum albumin) on the day of admission. HBV associated ACLF patients receive entecavir at the same time

ELIGIBILITY:
Inclusion Criteria:

1. age from 17ys to 70ys;
2. fale or femal;
3. ACLF, as deﬁned by the Asian Pacific Association for the Study of the Liver Working Party, is an acute hepatic insult manifested as jaundice (serum bilirubin ≥ 5 mg/dL) and coagulopathy[international normalized ratio (INR) ≥ 1.5 or prothrombin activity< 40%], with complications of ascites and/or encephalopathy within 4 wk in patients previously diagnosed or undiagnosed with chronic HBV associated liver disease and alcoholic liver

Exclusion Criteria:

1. super-infection or co-infection with hepatitis A, C, D, E,Epstein-Barr virus, cytomegalovirus, or human immunodeficiency virus;
2. a previous course immuno-modulator or cytotoxic/immunosuppressive therapy for chronic hepatitis within the prior 12 mo;
3. hepato-cellular carcinoma diagnosed by computed tomography or magnetic resonance imaging;
4. co-existence of any other serious medical illnesses or other liver diseases such as autoimmune hepatitis, drug-induced liver injury or Wilson's disease;
5. any concurrent evidence of sepsis;
6. malignant jaundice induced by obstructive jaundice and hemolytic jaundice;
7. prolonged prothrombin time due to blood system disease.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Survival rates | 12 weeks

SECONDARY OUTCOMES:
(Model of End Liver Disease,MELD) score | at 4 weeks; and at 12 weeks
(Sepsis-related Organ Failure Assessment,SOFA) score | at 4 weeks; and at 12 weeks
Total Bilirubin,TbiL | at 4 weeks; and at 12 weeks
incidence of complications;including infection, HRS | at 4 weeks; and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: jinhua hu, Dr. and PhD, Principal Investigator — Beijing; 302 Military Hospital
Locations (1):
- Beijing; 302 Military Hospital, Beijing, China

REFERENCES:
- [Derived] Tong J, Wang H, Xu X, Wan Z, Fang H, Chen J, Mu X, Liu Z, Chen J, Su H, Liu X, Li C, Huang X, Hu J. Granulocyte Colony-Stimulating Factor Accelerates the Recovery of Hepatitis B Virus-Related Acute-on-Chronic Liver Failure by Promoting M2-Like Transition of Monocytes. Front Immunol. 2022 May 16;13:885829. doi: 10.3389/fimmu.2022.885829. eCollection 2022. PMID 35651610